CLINICAL TRIAL: NCT03528759
Title: Streptococcus Pseudopneumoniae as an Emerging Respiratory Tract Pathogen at Assiut University Hospitals
Brief Title: Streptoccus Pseudopneumoniae atAssiut UniversityHospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Abdelfadeel, Principle Investigator, Assiut University
Other Study IDs: ZIS
Record Dates: First submitted 2018-03-26; First posted 2018-05-18 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2018-05

CONDITIONS: Pneumonia; Streptococcus Infection
MeSH Terms: conditions — Pneumonia; Streptococcal Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test:  — phenotypic and genotypic Method
  Other Names: Bile solubility test

SUMMARY:
Streptococcus pseudopneumoniae as suggested by DNA-DNA homology studies is recorded as a species of the Streptococcus mitis/oralis members of viridans group Streptococci; they have some similar features to the Streptococcus mitis/oralis members of viridans Streptococcus pneumoniae

DETAILED DESCRIPTION:
principle characteristics of Streptococcus. pseudopneumoniae are the lacking of pneumococcal capsule, bile insolubility, the indeterminate sensitivity Or resistance to optochin after incubation in Carbon dioxide (5%), while sensitivity to it after incubation in ambient air Streptococcus . pseudopneumoniae was firstly described in sputum samples of patients with lower respiratory tract infection, particularly those with Chronic Obstructive PulmonaryDiseases pseudopneumoniae is usually misidentified in our laboratories as we usually rely on optochin sensitivity testing with 5% Carbon dioxide detection of Streptococcus. pneumoniae and miss the incubation in ambient air which is the key point for identification of Streptococcus. pseudopneumoniae. Biochemical reactions are usually used to differentiate typical pneumoniae from Streptococc Streptococcus . pseudopneumoniae and other related Streptococci; several molecular techniques have also been used There are several polymerase chain reaction based assays that target specific pneumococcal virulence factors for the typical Streptococc Streptococcus . pneumoniae, such as autolysin A which is the major pneumococcal autolysin and the capsular polysaccharide biosynthesis gene A which is a conservedpneumococcal capsular polysaccharide gene , also aliB-like ORF2 (a gene that usually found in the capsular region of non-capsulated pneumococci; these genetic markers have been used to differentiate S. pneumoniae from other related species.

ELIGIBILITY:
Inclusion Criteria:

* All patients showing signs of respiratory tract infection

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sputum samples will be collected from all studied patients under complete aseptic condition. sputum specimens will be cultivated on 5% sheep blood agar, chocolate agar (Oxoid, UK.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-03 (Estimated)

PRIMARY OUTCOMES:
identification of Streptococcus. pseudopneumoniae | 1year
  Streptococcus will be identified by polymerase chain Reaction under complete aseptic condition

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Raddaoui A, Simoes AS, Baaboura R, Felix S, Achour W, Ben Othman T, Bejaoui M, Sa-Leao R, Ben Hassen A. Serotype Distribution, Antibiotic Resistance and Clonality of Streptococcus pneumoniae Isolated from Immunocompromised Patients in Tunisia. PLoS One. 2015 Oct 13;10(10):e0140390. doi: 10.1371/journal.pone.0140390. eCollection 2015. PMID 26461259
- [Result] Charalambous BM. Identifying divergent streptococcal strains using pherotype: implications for pathogen emergence and epidemiology. Future Microbiol. 2012 Dec;7(12):1349-54. doi: 10.2217/fmb.12.114. PMID 23231485
- [Result] Leung MH, Ling CL, Ciesielczuk H, Lockwood J, Thurston S, Charalambous BM, Gillespie SH. Streptococcus pseudopneumoniae identification by pherotype: a method to assist understanding of a potentially emerging or overlooked pathogen. J Clin Microbiol. 2012 May;50(5):1684-90. doi: 10.1128/JCM.00131-12. Epub 2012 Feb 29. PMID 22378913